CLINICAL TRIAL: NCT04094701
Title: Randomized Control Trial Evaluating Postoperative Opioid Demands Following Hip Arthroscopy
Brief Title: Hip Arthroscopy Postoperative Opioid Demands
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19071807
Record Dates: First submitted 2019-09-04; First posted 2019-09-19 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use; Pain; Femoral Acetabular Impingement; Labral Tear, Glenoid
MeSH Terms: conditions — Pain; Femoracetabular Impingement; Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Investigators propose two standardized prescribing patterns across all teams. The first would be the control postoperative prescribing pattern and the second would be the experimental opioid reduced prescribing pattern. Patients will not be informed if their postoperative prescriptions are part of the control or opioid reduced prescribing pattern. Of note, patients will be allowed to cross over from the opioid reduced experimental group to the standard of care control group if they have breakthrough pain following surgery.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group (Placebo Comparator): Control Group will receive the following pain medication regimen:
  - Norco (hydrocodone-acetaminophen) 5mg-325mg, 30 total pills
  The following non-opioid medications are standard of care at our practice following hip arthroscopy and, thus, will be prescribed to patients regardless of the group they are randomized to: aspirin (325 mg, two times daily for 30 days) and Indocin (75 mg extended release, one time daily for 10 days).
  Interventions: Other: Control Group Regimen
- Experimental Group - Opioid Reduced (Experimental): Experimental - opioid reduced: 50% less oxycodone relative to control group
  * Tylenol extra strength (1000 mg, three times daily for 10 days following surgery)
  * Gabapentin (300 mg at night for 10 days following surgery)
  * Norco (hydrocodone-acetaminophen) 5mg-325mg, 5 total pills
  The following non-opioid medications are standard of care at our practice following hip arthroscopy and, thus, will be prescribed to patients regardless of the group they are randomized to: aspirin (325 mg, two times daily for 30 days) and Indocin (75 mg extended release, one time daily for 10 days).
  Interventions: Other: Opioid reduced regimen

INTERVENTIONS:
Other: Control Group Regimen — Norco (hydrocodone-acetaminophen) 5mg-325mg, 30 total pills. This is the standard of care prescribing procedure for pain management after hip arthroscopy.
  Arms: Control Group
Other: Opioid reduced regimen — Tylenol extra strength (1000 mg, three times daily for 10 days following surgery), Gabapentin (300 mg at night for 10 days following surgery) and Norco (hydrocodone-acetaminophen) 5mg-325mg, 5 total pills
  Arms: Experimental Group - Opioid Reduced

SUMMARY:
This study will be a prospective, single-blinded, randomized controlled trial (RCT), investigating the influence of the number of opioid pills prescribed following primary hip arthroscopy. All patients who sign the consent form will be enrolled in the suited and randomized to one of the two treatment arms. The intervention group will receive 5 Norco pills, gabapentin (30 mg, once daily for 10 days following surgery), and Tylenol (1000 mg, three times daily for 10 days following surgery) while the control will receive the standard at our practice of 30 Norco pills.

DETAILED DESCRIPTION:
Follow-up will take place at 1, 3, 6, and 12 months postoperatively. Variables of interest will include postoperative patient pain scores (i.e. Visual Analog Scale or VAS), total morphine equivalents taken in the first 30 days after discharge, number of unused opioid pills, opioid disposal rates, and standard patient reported outcomes measures (PROMs) including hip disability and osteoarthritis outcome score (HOOS), Harris Hip score (HHS), VAS for pain, international hip outcome tool (iHOT-12), and Hip outcome score (HOS).

For the purpose of this study, the investigators propose two standardized prescribing patterns across all teams. The first would be the control postoperative prescribing pattern and the second would be the experimental opioid reduced prescribing pattern. Patients will not be informed if their postoperative prescriptions are part of the control or opioid reduced prescribing pattern. Of note, patients will be allowed to cross over from the opioid reduced experimental group to the standard of care control group if they have breakthrough pain following surgery.

Timeline of Events:

1. Following informed consent during the office visit when surgery is scheduled, all patients will be randomized to one of the postoperative pain management protocols, either the control or opioid reduced.
2. Subjects will proceed with hip arthroscopy, including appropriate treatment and documentation of concomitant injuries.
3. Over the course of the 1st month postoperatively, patients will complete a 30-day diary detailing which medications they took on each day and their daily average pain level (indicating whether physical therapy was performed). Data pertaining to prescription refills (I.e., number of refills, time to refill), number of left over pain medications, and disposal rates of opioid medications will also be recorded at these time points as well.
4. Patients will return for standard of care postoperative visits at 1, 3, 6, and 12 months postoperatively. Patients will be asked to complete PROM questionnaires at the 3, 6, and 12 month follow-up time points

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age 18-80 years
* English speaking
* Opioid naive patient (defined as not taking opioid pills within 6 weeks prior to surgery), confirmed by checking the Illinois Prescription monitoring program
* Primary hip arthroscopy
* Written and informed consent for study participation

Exclusion Criteria:

* Minors (<18 years of age)
* Opioid tolerant patients
* Revision surgery
* Prior infections of the operative joint
* History of active malignancy within the past 5 years
* Chronic pain conditions including low back pain, chronic pain syndrome, fibromyalgia
* History of alcohol or other substance use disorder
* Other disease states including rheumatologic conditions, diabetes mellitus, hypo/hyperthyroidism, depression, anxiety
* Grade IV chondral defects

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Pain Score | 1 month postoperatively
  Visual Analog Scale: unidimensional measure of pain intensity, which has been widely used in diverse adult populations. Score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Pain Score | 3 months postoperatively
  Visual Analog Scale: unidimensional measure of pain intensity, which has been widely used in diverse adult populations. Score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Pain Score | 6 months postoperatively
  Visual Analog Scale: unidimensional measure of pain intensity, which has been widely used in diverse adult populations. Score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Pain Score | 12 months postoperatively
  Visual Analog Scale: unidimensional measure of pain intensity, which has been widely used in diverse adult populations. Score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Total morphine equivalents taken | In the first 30 days after discharge
  Standardized reporting of amount of opioids taken
Number of unused opioid pills | In the first 30 days after discharge
  Pills not taken by patient
Opioid disposal rates | In the first 30 days after discharge
  Number of unused pills properly disposed of

SECONDARY OUTCOMES:
Hip disability and osteoarthritis outcome score | 1 month postoperatively
  assess the patient's opinion about their hip and associated problems and to evaluate symptoms and functional limitations related to the hip during a therapeutic process. The outcome score consists of 40 items assessing 5 subscales. The 5 separate patient-relevant dimensions are Pain (P), Symptoms (S), Activity limitations daily living (ADL), Function in sport and recreation (SP) and hip related quality of life (QOL).
  Pain (P) includes 10 items with a total score of 40 points, Symptoms (S) includes 5 items with a total score of 20, Activity limitations daily living (ADL) includes 17 items with a total score of 68 and finally Function in sport and recreation (SP) and hip related quality of life both include 4 items with a total score of 16 each. The outcome measure is transformed in a worst to best scale from 0 to 100, with 100 indicating no symptoms and 0 indicating extreme symptoms.
Hip disability and osteoarthritis outcome score | 3 months postoperatively
  assess the patient's opinion about their hip and associated problems and to evaluate symptoms and functional limitations related to the hip during a therapeutic process. The outcome score consists of 40 items assessing 5 subscales. The 5 separate patient-relevant dimensions are Pain (P), Symptoms (S), Activity limitations daily living (ADL), Function in sport and recreation (SP) and hip related quality of life (QOL).
  Pain (P) includes 10 items with a total score of 40 points, Symptoms (S) includes 5 items with a total score of 20, Activity limitations daily living (ADL) includes 17 items with a total score of 68 and finally Function in sport and recreation (SP) and hip related quality of life both include 4 items with a total score of 16 each. The outcome measure is transformed in a worst to best scale from 0 to 100, with 100 indicating no symptoms and 0 indicating extreme symptoms.
Hip disability and osteoarthritis outcome score | 6 months postoperatively
  assess the patient's opinion about their hip and associated problems and to evaluate symptoms and functional limitations related to the hip during a therapeutic process. The outcome score consists of 40 items assessing 5 subscales. The 5 separate patient-relevant dimensions are Pain (P), Symptoms (S), Activity limitations daily living (ADL), Function in sport and recreation (SP) and hip related quality of life (QOL).
  Pain (P) includes 10 items with a total score of 40 points, Symptoms (S) includes 5 items with a total score of 20, Activity limitations daily living (ADL) includes 17 items with a total score of 68 and finally Function in sport and recreation (SP) and hip related quality of life both include 4 items with a total score of 16 each. The outcome measure is transformed in a worst to best scale from 0 to 100, with 100 indicating no symptoms and 0 indicating extreme symptoms.
Hip disability and osteoarthritis outcome score | 12 months postoperatively
  assess the patient's opinion about their hip and associated problems and to evaluate symptoms and functional limitations related to the hip during a therapeutic process. The outcome score consists of 40 items assessing 5 subscales. The 5 separate patient-relevant dimensions are Pain (P), Symptoms (S), Activity limitations daily living (ADL), Function in sport and recreation (SP) and hip related quality of life (QOL).
  Pain (P) includes 10 items with a total score of 40 points, Symptoms (S) includes 5 items with a total score of 20, Activity limitations daily living (ADL) includes 17 items with a total score of 68 and finally Function in sport and recreation (SP) and hip related quality of life both include 4 items with a total score of 16 each. The outcome measure is transformed in a worst to best scale from 0 to 100, with 100 indicating no symptoms and 0 indicating extreme symptoms.
Harris Hip score | 1 month postoperatively
  gives a maximum of 100 points. Pain receives 44 points, function 47 points, range of motion 5 points, and deformity 4 points. Function is subdivided into activities of daily living (14 points) and gait (33 points). The higher the HHS, the less dysfunction.
Harris Hip score | 3 months postoperatively
  gives a maximum of 100 points. Pain receives 44 points, function 47 points, range of motion 5 points, and deformity 4 points. Function is subdivided into activities of daily living (14 points) and gait (33 points). The higher the HHS, the less dysfunction.
Harris Hip score | 6 months postoperatively
  gives a maximum of 100 points. Pain receives 44 points, function 47 points, range of motion 5 points, and deformity 4 points. Function is subdivided into activities of daily living (14 points) and gait (33 points). The higher the HHS, the less dysfunction.
Harris Hip score | 12 months postoperatively
  gives a maximum of 100 points. Pain receives 44 points, function 47 points, range of motion 5 points, and deformity 4 points. Function is subdivided into activities of daily living (14 points) and gait (33 points). The higher the HHS, the less dysfunction.
International hip outcome tool | 1 month postoperatively
  comprised of 33 questions. Patients are asked to place a mark on a Visual Analog Scale (VAS) line for each question, with "significantly impaired" on the far left and "no problems at all" on the far right. total score is then calculated as the mean of all VAS scores as measured in millimeters.
International hip outcome tool | 3 months postoperatively
  comprised of 33 questions. Patients are asked to place a mark on a Visual Analog Scale (VAS) line for each question, with "significantly impaired" on the far left and "no problems at all" on the far right. total score is then calculated as the mean of all VAS scores as measured in millimeters.
International hip outcome tool | 6 months postoperatively
  comprised of 33 questions. Patients are asked to place a mark on a Visual Analog Scale (VAS) line for each question, with "significantly impaired" on the far left and "no problems at all" on the far right. total score is then calculated as the mean of all VAS scores as measured in millimeters.
International hip outcome tool | 12 months postoperatively
  comprised of 33 questions. Patients are asked to place a mark on a Visual Analog Scale (VAS) line for each question, with "significantly impaired" on the far left and "no problems at all" on the far right. total score is then calculated as the mean of all VAS scores as measured in millimeters.
Hip outcome score | 1 month postoperatively
  questionnaire with a scoring system composed of 2 sub-scales. The Activities of Daily Living (ADL) sub-scale made of 19 items and a Sports sub-scale composed of 9 items. Both subscales are marked separately and 17 items from the Activities of daily living scale are scored from 0 to 4, with 0 being 'unable to do' and 4, 'no difficulty'. 'Not applicable' responses are also possible options. The total score is then multiplied by 4 to get the highest potential score which can be no greater than 68. An overall higher score from both of these sub-scales represents a greater level of function.
Hip outcome score | 3 months postoperatively
  questionnaire with a scoring system composed of 2 sub-scales. The Activities of Daily Living (ADL) sub-scale made of 19 items and a Sports sub-scale composed of 9 items. Both subscales are marked separately and 17 items from the Activities of daily living scale are scored from 0 to 4, with 0 being 'unable to do' and 4, 'no difficulty'. 'Not applicable' responses are also possible options. The total score is then multiplied by 4 to get the highest potential score which can be no greater than 68. An overall higher score from both of these sub-scales represents a greater level of function.
Hip outcome score | 6 months postoperatively
  questionnaire with a scoring system composed of 2 sub-scales. The Activities of Daily Living (ADL) sub-scale made of 19 items and a Sports sub-scale composed of 9 items. Both subscales are marked separately and 17 items from the Activities of daily living scale are scored from 0 to 4, with 0 being 'unable to do' and 4, 'no difficulty'. 'Not applicable' responses are also possible options. The total score is then multiplied by 4 to get the highest potential score which can be no greater than 68. An overall higher score from both of these sub-scales represents a greater level of function.
Hip outcome score | 12 months postoperatively
  questionnaire with a scoring system composed of 2 sub-scales. The Activities of Daily Living (ADL) sub-scale made of 19 items and a Sports sub-scale composed of 9 items. Both subscales are marked separately and 17 items from the Activities of daily living scale are scored from 0 to 4, with 0 being 'unable to do' and 4, 'no difficulty'. 'Not applicable' responses are also possible options. The total score is then multiplied by 4 to get the highest potential score which can be no greater than 68. An overall higher score from both of these sub-scales represents a greater level of function.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT04094701/Prot_SAP_000.pdf